CLINICAL TRIAL: NCT03811860
Title: Lithium Therapeutic Drug Monitoring; Once Daily Vs Twice Daily Dosing and the Impact of Kidney Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Virginia Fernandes, Clinical Practice Leader, Psychiatry, Mount Sinai Hospital, Canada
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-0289-A
Record Dates: First submitted 2019-01-10; First posted 2019-01-22 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Bipolar Disorder; Major Depressive Disorder
Keywords: lithium; pharmacokinetics; renal; kidney
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Once Daily Dosing (Active Comparator): In this arm of the study, participants receive the prescribed dose of lithium once daily at bedtime. After 4-6 days, a steady state lithium serum level and serum creatinine are taken, and they crossover to the other arm (twice daily dosing, if they have not already done so). Frequency of selected medication use is noted.
  Interventions: Diagnostic Test: Lithium level; Diagnostic Test: Serum Creatinine
- Twice Daily Dosing (Active Comparator): In this arm of the study, participants receive the prescribed dose of lithium divided into two daily doses. After 4-6 days a steady state lithium serum level and serum creatinine are taken, and they crossover to the other arm (once daily dosing, if they have not already done so).Frequency of selected medication use is noted.
  Interventions: Diagnostic Test: Lithium level; Diagnostic Test: Serum Creatinine

INTERVENTIONS:
Diagnostic Test: Lithium level — The level of lithium in the serum
Diagnostic Test: Serum Creatinine — The level of creatinine (as an indicator of kidney function, to approximate GFR) in the serum

SUMMARY:
Lithium is a mainstay in the treatment of bipolar disorder, and a frequently used adjunctive therapy for major depressive disorder. It is accepted practice to monitor lithium serum levels to monitor for efficacy and toxicity. However, studies on the difference in lithium levels between once and twice daily dosing, which also assess the impact of kidney function are scarce. The aim of this study is to quantify this pharmacokinetic difference, identify the impact of kidney function, in the context of estimating effects to inform feasibility and sample size needed for a larger well-powered study.

DETAILED DESCRIPTION:
Bipolar disorder is a chronic and recurring condition which causes functional impairment and increases lifetime suicide risk. Major depressive disorder likewise confers a high burden of illness on the affected population, and treatment is complicated by the fact 50-70% of patients treated with an initial agent do not achieve full remission of symptoms. There are numerous clinical practice guidelines which support the use of lithium as a first-line agent for bipolar disorder, and as an adjunctive therapy for major depressive disorder. Therapeutic ranges for lithium were established in the 1970s using multiple daily dose regimens, and therefore should not be directly applied to patients taking lithium once daily. The current standard of practice is to measure levels 12 hours post dose irrespective of once or twice daily administration. There is some evidence that lithium levels drawn 12 hours post dose are 10 - 26% higher when dosing lithium once daily compared to twice daily, however, the impact of kidney function on this difference has not been studied, and this difference in 12h post levels has not been confirmed via prospective data. Guidance on therapeutic drug monitoring (TDM) is vague with respect to interpretation of specific lithium blood levels for once daily dosing. Physicians may reduce a patient's dose based on a lithium level that is seemingly higher that target, even if the patient is clinically stable, putting the patient at risk for re-emergence of symptoms. Though it is known that lithium is excreted by the kidney, the impact of kidney function on the difference in lithium levels when dosed once daily compared to twice daily is not well understood. The results of this pilot study will help identify the impact of kidney function on lithium therapeutic drug monitoring in current practice, and potentially lead to a larger multi-center study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the inpatient psychiatry unit at Mount Sinai Hospital treated with lithium therapy (i.e. taking lithium before admission, or initiated on lithium therapy during hospitalization)

Exclusion Criteria:

* any patients who are currently pregnant
* patients taking lithium three times daily
* patients taking lithium with a specific dosing frequency for a documented clinical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Difference in lithium levels between once and twice daily dosing | once 2 steady state levels have been taken (4-12 days of intervention)
  The average of the difference in 12 hour post-dose serum level between the two dosing regimens (once daily and twice daily dosing)

SECONDARY OUTCOMES:
Correlation between renal function and difference in lithium level | once 2 steady state levels have been taken (4-12 days of intervention) and average creatinine clearance has been calculated
  Calculated correlation coefficient (r) for renal function (as estimated by calculation of creatinine clearance via Cockroft Gault) and mean percent change in serum lithium concentration when transitioning between once and twice daily dosing
Frequency of selected concurrent medication use | recorded upon enrollment, and every 4-6 days until study completion, up to 12 months
  Frequency of thiazide diuretic, loop diuretic, NSAID, and ACE inhibitor/ARB use

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no such plan